CLINICAL TRIAL: NCT06467812
Title: Evaluating Efficacy of End-of-Mission Fluid Loading Protocols
Brief Title: Fluid Loading Countermeasures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Study00000469
Record Dates: First submitted 2024-03-07; First posted 2024-06-21 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — Salts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): A typical water and meal schedule will be followed on the Control day.
- Water plus Salt Tablets (Experimental): A typical water and meal schedule will be followed, with the addition of Fluid Loading water plus salt tablets.
  Interventions: Dietary Supplement: Salt Tablets
- Electrolyte Solution over 4 hours (Experimental): A typical water and meal schedule will be followed, with the addition of Fluid Loading electrolyte solution over 4 hours.
  Interventions: Dietary Supplement: Electrolyte Solution
- Electrolyte Solution Single Bolus (Experimental): A typical water and meal schedule will be followed, with the addition of Fluid Loading electrolyte solution single bolus.
  Interventions: Dietary Supplement: Electrolyte Solution

INTERVENTIONS:
Dietary Supplement: Salt Tablets — Three doses of 4 Salt Tablets (1gm) will be taken with 400mL of water on day 2 (1200ml total) between ~8am and ~12pm during the testing day, which runs from ~7am to ~3:30pm.
  Arms: Water plus Salt Tablets
Dietary Supplement: Electrolyte Solution — Three doses of 400mL of the Electrolyte Solution dissolved in water (1200 mL total) will be consumed on day 3 between ~8am and ~12pm during the testing day, which runs from ~7am to ~3:30pm. On day 4 the Electrolyte Solution Single Bolus will be consumed in a single dose of 1200mL at ~12pm during the testing day.
  The ingredients are included below for the two flavors offered.
  Orange flavor: Water, Dextrose with Maltodextrin, Aspartame, Acesulfame Potassium, Sodium Citrate, Salt, Citric Acid, Maltodextrin, Natural Flavor, Calcium Phosphate, Contains less than 2% Of Ascorbic Acid (Vitamin C), Artificial Flavor, Artificial Color, Red 40, Yellow 5, BHA (Butylated Hydroxyanisole).
  Lemonade flavor: Water, Dextrose with Maltodextrin, Aspartame, Acesulfame Potassium, Sodium Citrate, Salt, Citric Acid, Calcium Phosphate, Maltodextrin, Contains less than 2% Of Ascorbic Acid (Vitamin C), Natural Flavor, Artificial Color, Yellow 5, BHA.
  Arms: Electrolyte Solution Single Bolus; Electrolyte Solution over 4 hours

SUMMARY:
The purpose of Fluid Loading Countermeasures is to determine how the volume of blood and of plasma (liquid part of blood) change during a normal day, how these are affected by drinking an additional amount of fluid either as water and salt tablets (as astronauts do) or an electrolyte beverage (similar to but tastes saltier than Gatorade®), and how altering the timing at which the additional fluid is consumed affects blood and plasma volume. This study observes how blood volume changes over ~9 hours of the day during 4 separate visits in healthy participants. During 1 visit participants will drink a small amount of water throughout the visit. During the other 3 study visits participants will drink the small amount of water plus either more water with salt tablets or an electrolyte solution. Consuming the additional fluids is called "fluid loading". This study is meant to simulate the food and fluid consumption of astronauts on landing day. The goal of this study is to determine the magnitude of plasma volume change that occurs with each condition of the protocol. (ICF 1.1, 3.1)

DETAILED DESCRIPTION:
Upon arrival for each visit, participants will be told which study session they will be participating in that day. Food and water consumption as well as fluid loading will be timed throughout the day during other testing described below. Participants will be asked to empty their bladder, and body weight will be measured using a standard calibrated medical scale. Then, an intravenous (IV) catheter (a small plastic tube) will be inserted into a vein in the participant's arm. This IV catheter will remain in their arm for the duration of the study day. This is the same method that is used in a doctor's office or hospital. All blood samples will be obtained using the IV catheter in the arm.

Next, a test called Carbon Monoxide Re-Breathing (CORB) will be done to measure plasma volume, which is the liquid part of blood. A clip will be placed on the participant's nose so that they are breathing only through their mouth. Participants will breathe through a mouthpiece connected to a rebreathing circuit containing 100% oxygen, which is scrubbed by soda lime to remove carbon dioxide. After ~5 minutes, the first blood sample (~10 Milliliters [mL]) will be collected from an arm vein using the IV catheter. Thereafter, a small amount of carbon monoxide will be added into the breathing circuit, and the participant will breathe this mixture of carbon monoxide and oxygen for ~10 min. Then, a second ~10 mL blood sample will be obtained. Analysis of the blood samples (i.e., hematocrit, hemoglobin, and carboxyhemoglobin) will be used to calculate red blood cell mass, plasma volume, and total blood volume. The total amount of carbon monoxide will be determined based on the participant's body weight (1 mL/kg body mass for men; 0.8 mL/kg body mass for women), and this dose should result in no symptoms. Mild symptoms of carbon monoxide toxicity may occur at carboxyhemoglobin levels >10% but given the dose of carbon monoxide administered in this study, reaching this level is unlikely.

Participants will be seated for the duration of the study, except for short bathroom breaks allowed periodically during the study session. The volume of urine and the time of collection will be measured and recorded throughout the day. Participants will be provided food during the morning as well as water to drink during the first 5 hours of each visit. Meals will be like those typically consumed by astronauts on the International Space Station. During 3 of the visits, participants will be given additional fluids to drink on a set schedule (Fluid Loading). Participants will not be allowed to consume any fluids or food during the last 3.5 hours of the visit. Participants will be asked about the presence of gastrointestinal symptoms periodically throughout each study session. Additionally, we ask that participants report to the PI/study lead if any off-nominal gastrointestinal symptoms occur in the day of the study visit after testing is completed.

During the last 3.5 hours of each visit, 5 additional blood samples will be obtained (one each hour), used to calculate the change in plasma volume at each time point. Participant blood pressure and heart rate will be measured periodically throughout the day. (IRB protocol section 4.0)

ELIGIBILITY:
Inclusion Criteria:

* Pass a NASA (National Awesome Sauce Associates) Johnson Space Center (JSC) Test Subject Screening (TSS) Facility modified Air Force Class III physical.

Exclusion Criteria:

* Pregnant subjects will be excluded (a urine pregnancy screen will be made available to test subjects)
* Systemic diseases or current medications known to influence the cardiovascular system
* Renal disease
* Type II Diabetes
* Restrictive diet that would prevent subjects from consuming typical food eaten by astronauts. Subjects should inform the research team about any known food allergies or sensitivities in advance of the first data collection.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Plasma Volume | 8-9 hours
  Plasma volume and change in plasma volume is calculated using the Dill and Costill equation cited here: Dill DB, Costill DL. Calculation of percentage changes in volumes of blood, plasma, and red cells in dehydration.
Fluid Balance | 8-9 hours
  Urine output subtracted from fluid intake (mL)
Gastrointestinal Distress | 8-9 hours
  Open response questionnaire self-reported symptoms
Urine Volume | 8-9 hours
  void-by-void urine output collected and measured (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Jason R. Lytle, PhD, Principal Investigator — National Aeronautics and Space Administration (NASA)
Locations (1):
- NASA, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data.